CLINICAL TRIAL: NCT01805310
Title: Pre-operative Bowel Preparation Prior to Minimally Invasive Sacral Colpopexy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halina M Zyczynski, MD (Other)
Responsible Party: Sponsor-Investigator, Halina M Zyczynski, MD, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO12020453
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Pelvic Organ Prolapse; Prolapse
Keywords: Pelvic organ prolapse; Prolapse; Cathartics; Mechanical bowel preparation
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse | interventions — Cathartics; magnesium citrate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bowel Preparation (Other): Women randomized to the bowel preparation arm will be instructed to consume 300cc of magnesium citrate no later than 3PM on preoperative day number one. They will also be placed on a clear liquid diet on preoperative day number one.
  Interventions: Other: Bowel preparation
- No bowel preparation (Other): Subjects randomized to no bowel preparation will be instructed to continue a regular diet on preoperative day number one.
  Interventions: Other: No bowel preparation

INTERVENTIONS:
Other: Bowel preparation — Subjects randomized to the mechanical bowel preparation arm will be instructed to consume 300cc of magnesium citrate no later than 3PM on preoperative day number one.
  Other Names: Magnesium citrate
  Arms: Bowel Preparation
Other: No bowel preparation — Subjects randomized to no bowel preparation will be instructed to continue a regular diet on preoperative day number one.
  Arms: No bowel preparation

SUMMARY:
Prior to surgery, gynecologists and urogynecologists have routinely prescribed preoperative mechanical bowel preparations in attempts to decrease the risk of infection, while also providing easier bowel manipulation and better visualization during surgery. However, many of these proposed benefits have never been proven, and usage of bowel preparations amongst surgeons remains highly variable. In both the general surgery and gynecology literature, researchers have begun to question the need for the vigorous preparations.

Aside from surgical visualization, urogynecologists have additional concerns about how bowel preparations may impact postoperative bowel function given up to half of women with pelvic floor disorders have baseline constipation and straining is known to impact surgical recovery. Many studies have addressed various postoperative fiber and laxative preparations in attempts to improve postoperative bowel-related symptomatology, but none have specifically looked at preoperative bowel preparations.

This study aims to determine if mechanical bowel preparation prior to minimally invasive sacral colpopexy affects patients' postoperative recovery, specifically related to bowel symptomatology; operative or post-operative complications; surgeons' perceptions of surgical difficulty directly attributed to the bowel; and post-operative return of normal bowel function.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years
* Planned laparoscopic or robotic-assisted sacral colpopexy

Exclusion Criteria:

* History of ulcerative colitis or Crohn's disease
* Prior large or small bowel resection
* Known diagnosis of gastroparesis
* Prior pelvic radiation
* History of abdominal or pelvic malignancy
* Planned concurrent bowel surgery/anal sphincteroplasty/ rectovaginal fistula repair
* Pregnancy
* Known allergic reactions to components of the study products
* Known renal insufficiency
* Non-English speaking as the primary study questionnaires are all currently in English only

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-02; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
PAC-SYM | 1 year
  Bowel symptomatology and bowel-related discomfort will be assessed with the Patient Assessment of Constipation Symptom Questionnaire (PAC-SYM), a 12-item questionnaire covering three domains: abdominal, rectal, and stool.

SECONDARY OUTCOMES:
Surgeon perception of bowel preparation | 1 year
  Immediately after completing the surgical case, surgeons will complete a 13-item surgeon questionnaire assessing degree of surgical difficulty and how it relates to the bowel. Operative time and consultations will also be recorded as objective measures of surgical difficulty.
Return of normal bowel function | 1 year
  A seven-day bowel diary will be obtained at baseline and in the first week after surgery. This log will include daily assessment of bowel frequency, type of bowel movement using the validated Bristol stool scale, degree of straining, and used of narcotics or laxatives.
Perioperative complications | 1 year
  Complications occurring in both groups will be recorded. These include, but are not limited to infections, bowel obstructions, visceral organ injuries, and readmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L Kantartzis, MD, Principal Investigator — University of Pittsburgh; Halina M Zyczynski, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States